CLINICAL TRIAL: NCT00184860
Title: The Value of CT-PET-MRI Image Fusion in Determining Radiation Treatment Volumes in Patients With a Squamous Cell Carcinoma of the Head-and-Neck Region, Who Are to be Treated With Definitive Radiotherapy
Brief Title: The Role of CT-PET-MRI Image Fusion in Determining Radiation Treatment Volumes of Head-and-Neck Cancer Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2004/153
Record Dates: First submitted 2005-09-12; First posted 2005-09-16 (Estimated); Last update posted 2007-04-27 (Estimated); Status verified 2007-04

CONDITIONS: Head and Neck Neoplasms
MeSH Terms: conditions — Head and Neck Neoplasms | interventions — Magnetic Resonance Spectroscopy

INTERVENTIONS:
Procedure: PET-scan, MRI-scan

SUMMARY:
Technical developments in radiation oncology are making it possible to deliver a prescribed radiation dose to radiation target volume with increasing accuracy.

Therefore it is becoming even more relevant to accurately define the radiation target volumes.

The current standard in defining radiation target volumes in patients with head-and-neck cancer is to combine physical examination data with a CT-scan in the treatment position.

The goal of this investigation is to analyse the rol of CT-PET-MRI image fusion in defining radiation target volumes.

ELIGIBILITY:
Inclusion Criteria:

Patients eligible for definitive radiotherapy with a Head and Neck Neoplasm (squamous cell carcinoma) in one of the following anatomical sites:

* oral cavity
* oropharynx
* hypopharynx
* larynx

Exclusion Criteria:

* age < 18 years
* pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80
Dates: Start 2003-06

CONTACTS AND LOCATIONS:
Overall Officials: Johannes H Kaanders, MD. PhD, Study Director — Radiation oncologist, Radboud University Nijmegen Medical Centre, Nijmegen, The Netherlands
Locations (1):
- Radboud University Nijmegen Medical Centre, Nijmegen, Gelderland, Netherlands